CLINICAL TRIAL: NCT03060694
Title: Screening Inpatients With Type 2 Diabetes for Nonalcoholic Fatty Liver Disease Using Controlled Attenuation Parameter and Liver Stiffness Measurements
Brief Title: Screening Diabetes Patients for NAFLD With Controlled Attenuation Parameter and Liver Stiffness Measurements
Status: Completed | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-16-045
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2017-03

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetes group: Patients in this group are recruited from both departments of endocrinology and gastroenterology. The diagnosis of diabetes is confirmed by medical history, using anti-diabetic medicines or laboratory tests.
  Interventions: Other: diabetes
- Non-diabetes group: Patients in this group are recruited from department of gastroenterology. The exclusion of diabetes is confirmed by medical history or laboratory tests.

INTERVENTIONS:
Other: diabetes — 1. a history of diabetes and using anti-diabetic medicines.
  2. fasting serum glucose level greater than 7.1mmol/L, or glycosylated hemoglobin percentage greater than 6.5%.
  Groups: Diabetes group

SUMMARY:
The purpose of this study is to compare the severity of NAFLD in diabetic patients to that in non-diabetic patients.

DETAILED DESCRIPTION:
1. Patient recruitment: eligible patients in the department of endocrinology and department of gastroenterology are encouraged to participate in this study.
2. Non-diabetic patients admitted to the department of gastroenterology for other gastroenterological diseases. If available, these patients' data will be collected as control groups. Each diabetic patient is matched with a non-diabetic patient by factors of age, gender and BMI.
3. Hepatic steatosis and fibrosis are diagnosed via controlled attenuation parameter (CAP) and liver stiffness measurement by FibroScan ®, respectively. According to the meta-analysis of individual patient data published recently, the CAP in dB/m will be adjusted by deducting 10dB/m from the CAP value for NAFLD/NASH patients, 10dB/m for diabetes patients and deducting/adding 4.4dB/m for each unit of BMI above/below 25kg/m2 over the range of 20-30kg/m2.
4. Regular laboratory tests are performed, including complete blood counts, liver function, renal function, coagulation function, glycosylated hemoglobin, lipid metabolism, urine albumin/creatinine ratio, 24-hour urine albumin.
5. Anthropometric data consists of height, weight, body mass index (the weight in kilograms divided by the square of the height in meters) and waist circumference.
6. The diabetic duration, diabetic complications, the grading of hypertension, and the history of anti-diabetic drugs are gathered from medical records.
7. The data are collected via EpiData software. They are input into computer twice by a single researcher to avoid typing errors.
8. Site monitoring and auditing: As a project for postgraduate thesis, this study is monitored and audited by the school of postgraduate. The research records will be checked in December, 2016, as a mid-term inspection
9. Statistical analysis plan: data are summarized and presented using appropriate descriptive statistics. The normality of continuous variables is assessed by skewness statistic and graphically by normal probability plot. Patients characteristics between those with and without diabetes, and in diabetes group, between those with and without elevated CAP are compared using independent t test, Chi-square, or Fisher's exact tests as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* type 2 diabetics

Exclusion Criteria:

* malignancy;
* severe cardiovascular complications;
* any history of chronic hepatitis (hepatitis B or C virus infection, autoimmune hepatitis, Wilson's disease, hemachromatosis);
* secondary causes of fatty liver ( glucocorticoids, amiodarone, tamoxifen);
* alcohol consuming (20grams per day for male, and 10 grams per day for female);
* any hints of type 1 diabetes ( ketoacidosis, ketonuria, using insulin within 1 year after diagnosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: inpatients in the department of endocrinology in Xinhua Hospital
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2016-09; Primary Completion 2017-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
controlled attenuation parameter; liver stiffness measure | one day

CONTACTS AND LOCATIONS:
Overall Officials: Zhengjie Xu, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiaotong Univerisity School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kwok R, Choi KC, Wong GL, Zhang Y, Chan HL, Luk AO, Shu SS, Chan AW, Yeung MW, Chan JC, Kong AP, Wong VW. Screening diabetic patients for non-alcoholic fatty liver disease with controlled attenuation parameter and liver stiffness measurements: a prospective cohort study. Gut. 2016 Aug;65(8):1359-68. doi: 10.1136/gutjnl-2015-309265. Epub 2015 Apr 14. PMID 25873639
- [Result] Karlas T, Petroff D, Sasso M, Fan JG, Mi YQ, de Ledinghen V, Kumar M, Lupsor-Platon M, Han KH, Cardoso AC, Ferraioli G, Chan WK, Wong VW, Myers RP, Chayama K, Friedrich-Rust M, Beaugrand M, Shen F, Hiriart JB, Sarin SK, Badea R, Jung KS, Marcellin P, Filice C, Mahadeva S, Wong GL, Crotty P, Masaki K, Bojunga J, Bedossa P, Keim V, Wiegand J. Individual patient data meta-analysis of controlled attenuation parameter (CAP) technology for assessing steatosis. J Hepatol. 2017 May;66(5):1022-1030. doi: 10.1016/j.jhep.2016.12.022. Epub 2016 Dec 28. PMID 28039099